CLINICAL TRIAL: NCT03561896
Title: Stereotactic Radiosurgery or Hypofractionated Image-Guided Radiotherapy to the Surgical Cavity After Resection of Brain Metastases: a Multicenter, Single Arm, Open-label, Phase II Trial
Brief Title: Hypofractionated Brain Radiationcavity
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Oncology Institute of Southern Switzerland (Other)
Responsible Party: Principal Investigator, Gianfranco Angelo Pesce, MD, Oncology Institute of Southern Switzerland
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IOSI-RTO-001
Record Dates: First submitted 2017-01-19; First posted 2018-06-19 (Actual); Last update posted 2024-07-17 (Actual); Status verified 2024-07

CONDITIONS: Brain Metastases, Adult; Cancer Brain
Keywords: Radation therapy; sterotactic radiosurgery; quality of life; solid cancer; palliation; neurologic functionning
MeSH Terms: conditions — Brain Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- IGRT (Experimental): Image-Guided Hypofractionated Stereotactic Radiation Therapy (IGRT) of the resection cavity
  Interventions: Radiation: IGRT
- SRS (Experimental): Stereotactic Radiosurgery of the resection cavity (SRS)
  Interventions: Radiation: SRS

INTERVENTIONS:
Radiation: IGRT — Image-Guided Radiation Therapy
  Arms: IGRT
Radiation: SRS — stereotactic radiation therapy
  Arms: SRS

SUMMARY:
Stereotactic radiosurgery or hypofractionated radiotherapy of the resection cavity after metastasectomy in cancer patients with brain metastases

DETAILED DESCRIPTION:
Patients with limited number of brain metastases from solid tumors are at high risk of local recurrence after surgical removal of the tumor mass. The standard Whole-brain radiotherapy (WBRT) demonstrated to reduce the risk of recurrence without improving survival. At the same time WBRT have substantial acute and late toxicity. Preliminary experiences with Stereotactic radiosurgery or hypofractionated radiotherapy of the resection cavity indicate promising local control and good tolerance. This attitude was only partially explored in prospective trials. In this research patients with limited number of brain metastases and controlled systemic disease will be treated, with such a stereotactic irradiation, at the same time with evaluation of the local control (Primary endpoint) by repeated MRI and of quality of life, neurologic functionning (with a battery of thsts, e.g. MMSE, QLQ-C30, EORTC BN-20) as well as overall survival as secondary endpoints.

ELIGIBILITY:
Inclusion criteria:

* Patient underwent surgery for single brain metastasis arising from solid neoplasia (lung, breast, melanoma, kidney, colorectal), with initial histological diagnosis, or selected cases with a resected lesion and a further non-resected lesion (from 1 to 2 lesions), treatable with SRS / IGRT of the surgical cavity
* Patient ≥ 18 years
* Willngness to participate in the study, written informed consent
* Performance Status according to WHO 0-I
* Good general conditions and organ function
* Newly diagnosed chemotherapy-naïve disease or controlled systemic disease
* Good bone marrow, renal and hepatic function
* Stable steroid dose or reduced for at least 5 days

Exclusion Criteria:

* History of previous brain irradiation
* Pregnancy or breastfeeding
* Histological diagnosis other than lung, breast, melanoma, kidney and colorectal malignancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 56 (Actual)
Dates: Start 2015-01 (Actual); Primary Completion 2024-06-18 (Actual); Study Completion 2024-06-18 (Actual)

PRIMARY OUTCOMES:
Relapse rate | 1 year
  Evaluate the recurrence probability in the surgical cavity after radiotherapy

SECONDARY OUTCOMES:
Overall survival | 1 year
  The proportion of surviving patients at 1 year
Time to systemic progression | 1 year
  The proportion of patients with progression of disease in any location other than the brain, according to CTCAE Criteria
Time to neurological progression | 1 year
  Time to neurological deterioration (objective neurological examination and MMSE)
Quality of life assessment | 1 year
  Evaluation of the quality of life through questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Gianfranco A Pesce, MD, Principal Investigator — IOSI, Bellinzona, Switzerland
Locations (6):
- Switzerland (6):
  - Oncology Institute of Southern Switzerland (IOSI), Bellinzona, Canton Ticino
  - Universitätsspital Basel, Basel
  - Inselspital, Bern
  - Kantonsspital Winterthur, Winterthur
  - Klinik Hirslanden, Zurich
  - University Hospital Zurich (USZ), Zurich

IPD SHARING:
Plan to Share IPD: Undecided